CLINICAL TRIAL: NCT06369649
Title: Effect of Coolsense and Buzzy Use on Pain Score and Anxiety Level During Insulin Injection Application in Children With Type 1 Diabetes Mellitus
Brief Title: Coolsense and Buzzy Use on Pain Score and Anxiety Level During Insulin Injection Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Mine Nur Temuçin, research assistant, faculty of health science, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: COOLSENSE-1
Record Dates: First submitted 2024-02-05; First posted 2024-04-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Injection Fear; Injection Site Coldness; Pain; Type 1 Diabetes Mellitus; Pediatric Disease; Nurse's Role
Keywords: Injection fear; Injection pain; Pain; Type 1 Diabetes Mellitus; Pediatric Disease; Nursing
MeSH Terms: conditions — Iatrophobia; Pain; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinding (participants) will be used in the research and the researchers will not have information about the other group.
  While applying both scales, care will be taken to ensure that children, parents and observers do not see each other's evaluations and are not influenced by each other. In this way, the child, parent and independent observer will score blindly before and after the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coolsense (Experimental): For children in this group, the standard approach of the clinic will be applied first. The researcher will apply scales to the child before the procedure, the Child-Parent Information Form to the parents, and the child, parent and independent observer before and after the procedure. The patient's physiological parameters will be recorded by the nurse performing the procedure before, during and after the procedure. The device, which is removed from the freezer just before the injection, will be applied by the researcher to the skin surface where the procedure will be performed for approximately 5-10 seconds before the injection, and then the injection will be performed.
  Interventions: Device: Coolsense and Buzzy
- Buzzy (Experimental): For children in this group, the standard approach of the clinic will be applied first. The researcher will apply scales to the child before the procedure, the Child-Parent Information Form to the parents, and the child, parent and independent observer before and after the procedure. The patient's physiological parameters will be recorded by the nurse performing the procedure before, during and after the procedure. The device, which will be removed from the freezer just before the injection, will be placed by the researcher in contact with the skin, 3 to 5 cm above the injection site. Buzzy will be started 30-60 seconds before the process and will continue until the end of the process.
  Interventions: Device: Coolsense and Buzzy
- Control (No Intervention): For children in this group, the standard approach of the clinic will be applied first. The researcher will apply scales to the child before the procedure, the Child-Parent Information Form to the parents, and the child, parent and independent observer before and after the procedure. The patient's physiological parameters will be recorded by the nurse performing the procedure before, during and after the procedure.

INTERVENTIONS:
Device: Coolsense and Buzzy — Before the procedure, the independent observer, parent and child will be informed by the researcher about the method that will be used in the selected group and the scales that they will score. For children and parents in each group, a standard approach will be applied. Single blinding (participants) will be used in the research and the researchers will not have information about the other group. Cold application will be applied to children in group number one (Coolsense group). Coolsense, which does not contain any chemicals, provides cold application with the metal piece on its tip. In group number two (Buzzy group), vibration and cold application will be applied to the children. Buzzy is a handheld device with a bee-shaped motor that creates a small cold pad and vibration in the area in contact with the skin surface. Group number three (control group) will continue the standard procedure of the clinic and no different application or approach will be applied.
  Other Names: Buzzy; Coolsense
  Arms: Buzzy; Coolsense

SUMMARY:
This study aims to determine the effect of using Coolsense, which is created using the proven effect of cold application during insulin injection, and Buzzy, which is a combination of vibration and cold application, in reducing pain and anxiety in children diagnosed with Type 1 diabetes mellitus.This randomized controlled clinical study is planned to be conducted between 05.2024-12.2025 with 147 participants between the ages of 6-12. Participants will be divided into three groups according to the randomization method: buzzy group (n = 49), coolsense group (n = 49) and control group (n = 49). Participants in the Coolsense group will receive a cold application using the coolsense device for 5 seconds before the injection. Participants in the Buzzy group will be subjected to vibration and cold application 30-60 seconds before the procedure. Participants in the control group will continue the clinic's standard procedure. Changes in participants' pain score and fear level, heart rate, blood pressure, respiratory rate and oxygen saturation will be measured at three time points: immediately before and after the procedure. Data descriptive information form, application registration form, Facial Expressions Pain Scale (FPS-R) and Child Fear Scale (CFS) will be used. The collected data will be analyzed using SPSS 15 software. The main questions it aims to answer:

* Does buzzy and coolsense application have an effect the pain score of children during the insülin injection?
* Does buzzy and coolsense application have an effect the fear score of children during the insülin injection?

DETAILED DESCRIPTION:
Children between the ages of 6-10, who is diagnosed at least 2 weeks ago, will be included in the study.Patients with intellectual or neurological disabilities, Raynaud syndrome or sickle cell anemia will excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Being an inpatient in the Pediatric Endocrinology Service
* Having a diagnosis of Type 1 Diabetes Mellitus (no more than 6 months have passed since the diagnosis) receiving insulin therapy
* Being in the 6-10 age group.
* Having no pain before the application (getting 0 points on the pain scale).
* Blood sugar level above 80 mg/dl
* Having parental permission
* The child's willingness to participate in the research
* Not having used any medication that would have an analgesic effect in the last 24 hours before application.
* The child does not have a mental or neurological disability
* Not having any disease that causes sensitivity to cold, such as Reynaud's syndrome or sickle cell anemia.
* The child must be conscious and have no communication problems
* The child and the parent must be able to speak Turkish

Exclusion Criteria:

* Being younger than 6 years old and older than 12 years old
* Not having a diagnosis of Type 1 Diabetes
* Presence of pain before application
* Blood glucose level should be below 80 mg/dl before application
* The person or the parent does not agree to participate in the research.
* Having a disease that causes chronic pain
* Presence of any incision or scar tissue in the area to be injected

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale- Revised (FPS-R) | just before injection, just after injection
  It consists of facial expressions to evaluate pain intensity and is used in children aged four years and above. The scale consists of six simplified facial expressions that indicate the intensity of pain at increasing levels from 0 to 10 (0-2-4-6-8-10). In the scale, the child is asked to show the facial expression that best describes the intensity of pain. 0 means no pain, 10 means no pain indicates severe pain.
Children's Fear Scale (CFS) | just before injection, just after injection
  The scale used to evaluate the level of anxiety in children is a visual measurement tool that consists of five drawn facial expressions ranging from neutral expression (0 = no anxiety) to scared face (4 = severe anxiety) and receives a score of 0-4 points. As the score obtained from the scale increases, the severity of anxiety increases, and as the score decreases, anxiety decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Nur TEMUÇİN, MSc, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erdogan B, Aytekin Ozdemir A. The Effect of Three Different Methods on Venipuncture Pain and Anxiety in Children: Distraction Cards, Virtual Reality, and Buzzy(R) (Randomized Controlled Trial). J Pediatr Nurs. 2021 May-Jun;58:e54-e62. doi: 10.1016/j.pedn.2021.01.001. Epub 2021 Jan 21. PMID 33485746
- [Result] Susam V, Friedel M, Basile P, Ferri P, Bonetti L. Efficacy of the Buzzy System for pain relief during venipuncture in children: a randomized controlled trial. Acta Biomed. 2018 Jul 18;89(6-S):6-16. doi: 10.23750/abm.v89i6-S.7378. PMID 30038198
- [Result] Xess PA, Sarna R, Sethi S, Chauhan R, Meena SC, Saini V, Luthra A, Singh N. Effect of CoolSense and EMLA Cream on Pain During Intravenous Cannulation in Pediatric Population: A Randomized, Controlled Trial. Indian J Pediatr. 2024 Feb;91(2):119-124. doi: 10.1007/s12098-022-04233-w. Epub 2022 Jun 29. PMID 35767175